CLINICAL TRIAL: NCT03401424
Title: The RCT Study of Two Surgical Biliary-enteric Reconstruction Minimally Invasive Treatment of Bile Duct Dilatation
Brief Title: Comparison of Two Kinds of Biliary Intestinal Reconstruction in Cholangiectasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shuguo Zheng, MD, Professor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SWHZSG008; Zhengshuguo (Registry Identifier: Zhengshuguo)
Record Dates: First submitted 2017-12-28; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Postcholecystectomy Syndrome
Keywords: congenital cyst of common bile duct; Biliary enteric anastomosis
MeSH Terms: conditions — Postcholecystectomy Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- improved Warren-type style (Experimental): Minimally invasive treatment improved Warren-type cholangiocarcinoma reconstruction is easy
  Interventions: Procedure: improved Warren-type style
- Roux-en-Y style (Active Comparator): Early open cholecystectomy reconstruction surgery using Roux-en-Y style
  Interventions: Procedure: Roux-en-Y style

INTERVENTIONS:
Procedure: improved Warren-type style — Select 60 cases of biliary dilatation in patients undergoing laparoscopic cyst excision plus modified Warren cholangiobiliary reconstruction.
  Arms: improved Warren-type style
Procedure: Roux-en-Y style — Select 60 cases of biliary dilatation in patients undergoing laparoscopic cyst excision Roux-en-Y cholangiobiliary reconstruction.
  Arms: Roux-en-Y style

SUMMARY:
To observe and compare the short-term and long-term effects of different biliary and intestinal reconstruction methods for the treatment of congenital cystic dilatation of bile duct .

DETAILED DESCRIPTION:
The purpose of the study： length of operation time, postoperative intestinal function recovery time as the main index, application prospective clinical study to observe the differences were followed by two different laparoscopic biliary intestinal kiss the short-term and long-term effect of the treatment of congenital cystic dilatation of the bile duct, provide a higher level of evidence based medicine dilatation of patients for congenital bile duct cysts. The choice of second is based on the study, effective, objective evaluation of different laparoscopic biliary enteric reconstruction for the treatment of congenital cystic dilatation of the bile duct is feasible, clear surgical indications, contraindications and summarized the technical points, establish guidelines for clinical diagnosis and treatment of congenital cystic dilation of the bile duct disease.

ELIGIBILITY:
Inclusion Criteria:

1. gender, age 5-70 years old (the disease can occur at any age, but in 80% cases of childhood onset, such as children's height and weight of endoscopic treatment for the standard, by parents as guardians into the group);
2. preoperative congenital cystic dilatation of the bile duct (I, II, IV) clear diagnosis; preoperative assessment of liver function
3. : Child-Pugh = B;
4. bile duct without canceration;
5. recurrent cholangitis, biliary calculi in the biliary tract infection was controlled in acute pancreatitis; control of inflammation;
6. the treatment of choledochal cyst, without any surgical treatment;
7. the general condition of the patient, heart and lung function can tolerate surgery, no absolute contraindication abdominal laparoscopic operation;
8. voluntarily participated in the study, informed consent.

Exclusion Criteria:

1. congenital cystic dilatation of the bile duct of III type, V type (III type feasible endoscope end of bile duct duodenal sphincterotomy, V type partial resection of the liver);
2. patients who cannot tolerate pneumoperitoneum or serious abdominal adhesions, unable to carry out laparoscopic surgery;
3. bad general condition or heart pulmonary dysfunction cannot tolerate surgery;
4. severe cholestatic cirrhosis, severe portal hypertension;
5. high risk patients with general anesthesia.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
operation time | 2 years
  Two surgical methods operation time

CONTACTS AND LOCATIONS:
Overall Officials: Shuguo Zheng, Study Director — Shuguo Zheng, MD Study Director Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No